CLINICAL TRIAL: NCT00159835
Title: Atorvastatin Compared With Simvastatin In The Prevention of CHD Morbidity And Mortality In Patients With CHD
Brief Title: Atorvastatin Versus Simvastatin In The Prevention Of Coronary Heart Disease (CHD) In Patients With Known CHD
Acronym: IDEAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATV-N-98-001; A2581145
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Atorvastatin; Simvastatin

INTERVENTIONS:
Drug: atorvastatin
Drug: simvastatin

SUMMARY:
To investigate whether a long-term strategy to lower LDL cholesterol with atorvastatin as much as possible will improve prognosis in CHD patients compared with a strategy reflecting current best clinical practice with simvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Previous myocardial infarction

Exclusion Criteria:

* Women who are breast feeding or are pregnant

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8600
Dates: Start 1999-02; Study Completion 2005-03

PRIMARY OUTCOMES:
Time to of a major coronary event: 1) non-fatal acute myocardial infarction 2) coronary death 3) resuscitated cardiac arrest

SECONDARY OUTCOMES:
1) Time to any CHD event, 2) Time to Hospitalization with primary diagnosis of CHF, 3) Time to Cerbrovascular Event, 4) Time to PAD, 5) Time to any CV event and 6) All Cause Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (161):
- Denmark (28):
  - Pfizer Investigational Site, Arhus C
  - Pfizer Investigational Site, Copenhagen
  - Pfizer Investigational Site, Elsinore
  - Pfizer Investigational Site, Esbjerg
  - Pfizer Investigational Site, Fredericia
  - Pfizer Investigational Site, Frederiksberg
  - Pfizer Investigational Site, Frederikssund
  - Pfizer Investigational Site, Grenå
  - Pfizer Investigational Site, Hjørring
  - Pfizer Investigational Site, Holbak
  - Pfizer Investigational Site, Holstebro
  - Pfizer Investigational Site, Hvidovre
  - Pfizer Investigational Site, Kabenhavn S
  - Pfizer Investigational Site, Kalundborg
  - Pfizer Investigational Site, KÃ¸benhavn NV
  - Pfizer Investigational Site, Kobenhavn K
  - Pfizer Investigational Site, København NV
  - Pfizer Investigational Site, Køge
  - Pfizer Investigational Site, Middelfart
  - Pfizer Investigational Site, Nykøbing Falster
  - Pfizer Investigational Site, Næstved
  - Pfizer Investigational Site, Odder
  - Pfizer Investigational Site, Randers
  - Pfizer Investigational Site, Roskilde
  - Pfizer Investigational Site, Silkeborg
  - Pfizer Investigational Site, Skive
  - Pfizer Investigational Site, Slagelse
  - Pfizer Investigational Site, Svendborg
- Finland (16):
  - Pfizer Investigational Site, Ekenäs
  - Pfizer Investigational Site, Heinola
  - Pfizer Investigational Site, Helsinki
  - Pfizer Investigational Site, Joensuu
  - Pfizer Investigational Site, Jyväskylä
  - Pfizer Investigational Site, Kerava
  - Pfizer Investigational Site, Kuopio
  - Pfizer Investigational Site, Lahti
  - Pfizer Investigational Site, Lappeenranta
  - Pfizer Investigational Site, Lohja
  - Pfizer Investigational Site, Mikkeli
  - Pfizer Investigational Site, Rauma
  - Pfizer Investigational Site, Salo
  - Pfizer Investigational Site, Siaraalamaki
  - Pfizer Investigational Site, Tampere
  - Pfizer Investigational Site, Vantaa
- Pfizer Investigational Site, Reykjavik, Iceland
- Netherlands (23):
  - Pfizer Investigational Site, 's-Hertogenbosch
  - Pfizer Investigational Site, Alkmaar
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, Assen
  - Pfizer Investigational Site, Breda
  - Pfizer Investigational Site, Capelle aan den IJssel
  - Pfizer Investigational Site, Delft
  - Pfizer Investigational Site, Deventer
  - Pfizer Investigational Site, Ede
  - Pfizer Investigational Site, Eindhoven
  - Pfizer Investigational Site, Enschede
  - Pfizer Investigational Site, Goes
  - Pfizer Investigational Site, Groningen
  - Pfizer Investigational Site, Hoorn
  - Pfizer Investigational Site, Nijmegen
  - Pfizer Investigational Site, Oss
  - Pfizer Investigational Site, Rotterdam
  - Pfizer Investigational Site, Tilburg
  - Pfizer Investigational Site, Tilurg
  - Pfizer Investigational Site, Utrecht
  - Pfizer Investigational Site, Weert
  - Pfizer Investigational Site, Zwijndrecht
  - Pfizer Investigational Site, Zwolle
- Norway (41):
  - Pfizer Investigational Site, Ålesund
  - Pfizer Investigational Site, Bergen
  - Pfizer Investigational Site, Bodø
  - Pfizer Investigational Site, Flekkefjord
  - Pfizer Investigational Site, Førde
  - Pfizer Investigational Site, Hammerfest
  - Pfizer Investigational Site, Haugesund
  - Pfizer Investigational Site, HobÃ¸l
  - Pfizer Investigational Site, Jessheim
  - Pfizer Investigational Site, Karasjok
  - Pfizer Investigational Site, Kongsberg
  - Pfizer Investigational Site, Kongsvinger
  - Pfizer Investigational Site, Kragerø
  - Pfizer Investigational Site, Kristiansand
  - Pfizer Investigational Site, Kristiansund N
  - Pfizer Investigational Site, Larvik
  - Pfizer Investigational Site, Levanger
  - Pfizer Investigational Site, Lillestom
  - Pfizer Investigational Site, Lorenskog
  - Pfizer Investigational Site, Mo i Rana
  - Pfizer Investigational Site, Molde
  - Pfizer Investigational Site, MosjÃ¸en
  - Pfizer Investigational Site, Moss
  - Pfizer Investigational Site, Mysen
  - Pfizer Investigational Site, Nesttun
  - Pfizer Investigational Site, Notodden
  - Pfizer Investigational Site, Odda
  - Pfizer Investigational Site, Oslo
  - Pfizer Investigational Site, Paradis
  - Pfizer Investigational Site, Porsgrunn
  - Pfizer Investigational Site, Rud
  - Pfizer Investigational Site, Sandvika
  - Pfizer Investigational Site, Skedsmokorset
  - Pfizer Investigational Site, Ski
  - Pfizer Investigational Site, Stavanger
  - Pfizer Investigational Site, Stord
  - Pfizer Investigational Site, Tansberg
  - Pfizer Investigational Site, Trondheim
  - Pfizer Investigational Site, Tynset
  - Pfizer Investigational Site, Tønsberg
  - Pfizer Investigational Site, Volda
- Sweden (51):
  - Pfizer Investigational Site, Alingsås
  - Pfizer Investigational Site, Ängelholm
  - Pfizer Investigational Site, Bålsta
  - Pfizer Investigational Site, Borås
  - Pfizer Investigational Site, Eksjö
  - Pfizer Investigational Site, Eskilstuna
  - Pfizer Investigational Site, Fagersta
  - Pfizer Investigational Site, Falköping
  - Pfizer Investigational Site, Falun
  - Pfizer Investigational Site, Finspång
  - Pfizer Investigational Site, Gateborg
  - Pfizer Investigational Site, Gävle
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Grästorp
  - Pfizer Investigational Site, Halmstad
  - Pfizer Investigational Site, Hässleholm
  - Pfizer Investigational Site, Helsingborg
  - Pfizer Investigational Site, Hudiksvall
  - Pfizer Investigational Site, Jönköping
  - Pfizer Investigational Site, Kalmar
  - Pfizer Investigational Site, Karlshamn
  - Pfizer Investigational Site, Karlskoga
  - Pfizer Investigational Site, Karlskrona
  - Pfizer Investigational Site, Karlstad
  - Pfizer Investigational Site, Katarineholm
  - Pfizer Investigational Site, Köping
  - Pfizer Investigational Site, Kristinehamn
  - Pfizer Investigational Site, Lidköping
  - Pfizer Investigational Site, Linka Ping
  - Pfizer Investigational Site, Ljungby
  - Pfizer Investigational Site, Ludvika
  - Pfizer Investigational Site, Luleå
  - Pfizer Investigational Site, Lycksele
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Mariestad
  - Pfizer Investigational Site, Motala
  - Pfizer Investigational Site, Mölndal
  - Pfizer Investigational Site, Norrköping
  - Pfizer Investigational Site, Sala
  - Pfizer Investigational Site, Sandviken
  - Pfizer Investigational Site, Skellefteå
  - Pfizer Investigational Site, Skene
  - Pfizer Investigational Site, Skövde
  - Pfizer Investigational Site, Södertälje
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Strömstad
  - Pfizer Investigational Site, Uddevalla
  - Pfizer Investigational Site, Umeå
  - Pfizer Investigational Site, Varberg
  - Pfizer Investigational Site, VÃ¤nersborg
  - Pfizer Investigational Site, Västervik
- Pfizer Investigational Site

REFERENCES:
- [Result] Pedersen TR, Faergeman O, Kastelein JJ, Olsson AG, Tikkanen MJ, Holme I, Larsen ML, Bendiksen FS, Lindahl C, Szarek M, Tsai J; Incremental Decrease in End Points Through Aggressive Lipid Lowering (IDEAL) Study Group. High-dose atorvastatin vs usual-dose simvastatin for secondary prevention after myocardial infarction: the IDEAL study: a randomized controlled trial. JAMA. 2005 Nov 16;294(19):2437-45. doi: 10.1001/jama.294.19.2437. PMID 16287954
- [Derived] Tunnicliffe DJ, Palmer SC, Cashmore BA, Saglimbene VM, Krishnasamy R, Lambert K, Johnson DW, Craig JC, Strippoli GF. HMG CoA reductase inhibitors (statins) for people with chronic kidney disease not requiring dialysis. Cochrane Database Syst Rev. 2023 Nov 29;11(11):CD007784. doi: 10.1002/14651858.CD007784.pub3. PMID 38018702
- [Derived] Ports WC, Fayyad R, DeMicco DA, Laskey R, Wolk R. Effectiveness of Lipid-Lowering Statin Therapy in Patients With and Without Psoriasis. Clin Drug Investig. 2017 Aug;37(8):775-785. doi: 10.1007/s40261-017-0533-0. PMID 28573499
- [Derived] Stam-Slob MC, van der Graaf Y, Greving JP, Dorresteijn JA, Visseren FL. Cost-Effectiveness of Intensifying Lipid-Lowering Therapy With Statins Based on Individual Absolute Benefit in Coronary Artery Disease Patients. J Am Heart Assoc. 2017 Feb 18;6(2):e004648. doi: 10.1161/JAHA.116.004648. PMID 28214794
- [Derived] Deedwania PC, Pedersen TR, DeMicco DA, Breazna A, Betteridge DJ, Hitman GA, Durrington P, Neil A; TNT, CARDS and IDEAL Steering Committees and Investigators. Differing predictive relationships between baseline LDL-C, systolic blood pressure, and cardiovascular outcomes. Int J Cardiol. 2016 Nov 1;222:548-556. doi: 10.1016/j.ijcard.2016.07.201. Epub 2016 Jul 30. PMID 27513651
- [Derived] Stoekenbroek RM, Boekholdt SM, Fayyad R, Laskey R, Tikkanen MJ, Pedersen TR, Hovingh GK; Incremental Decrease in End Points Through Aggressive Lipid Lowering Study Group. High-dose atorvastatin is superior to moderate-dose simvastatin in preventing peripheral arterial disease. Heart. 2015 Mar;101(5):356-62. doi: 10.1136/heartjnl-2014-306906. Epub 2015 Jan 16. PMID 25595417
- [Derived] Dorresteijn JA, Boekholdt SM, van der Graaf Y, Kastelein JJ, LaRosa JC, Pedersen TR, DeMicco DA, Ridker PM, Cook NR, Visseren FL. High-dose statin therapy in patients with stable coronary artery disease: treating the right patients based on individualized prediction of treatment effect. Circulation. 2013 Jun 25;127(25):2485-93. doi: 10.1161/CIRCULATIONAHA.112.000712. Epub 2013 May 14. PMID 23674398
- [Derived] Semb AG, Kvien TK, DeMicco DA, Fayyad R, Wun CC, LaRosa JC, Betteridge J, Pedersen TR, Holme I. Effect of intensive lipid-lowering therapy on cardiovascular outcome in patients with and those without inflammatory joint disease. Arthritis Rheum. 2012 Sep;64(9):2836-46. doi: 10.1002/art.34524. PMID 22576673
- [Derived] Hyde CL, Macinnes A, Sanders FA, Thompson JF, Mazzarella RA, Faergeman O, van Wijk DF, Wood L, Lira M, Paciga SA. Genetic association of the CCR5 region with lipid levels in at-risk cardiovascular patients. Circ Cardiovasc Genet. 2010 Apr;3(2):162-8. doi: 10.1161/CIRCGENETICS.109.897793. Epub 2010 Feb 3. PMID 20130232